CLINICAL TRIAL: NCT02477059
Title: Double-blind, Randomized, Placebo-controlled Trial Evaluating the Effect of Two Infusions Four Weeks Apart of Interleukin-6-Receptor Inhibitor (Tocilizumab) on Pain Relief in Patients With Severe Osteoarthritis of the Hand Refractory to Usual Treatment
Brief Title: Effect of the Interleukin-6 Receptor Antagonist Tocilizumab in Patients With Hand Osteoarthritis
Acronym: TIDOA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P120206
Record Dates: First submitted 2015-06-10; First posted 2015-06-22 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Hand Osteoarthritis
Keywords: Hand OA; Tocilizumab; Osteoarthritis; Interleukin-6
MeSH Terms: conditions — Osteoarthritis | interventions — tocilizumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tocilizumab (Experimental): 2 infusions four weeks apart
  Interventions: Drug: tocilizumab
- saline solution (Placebo Comparator): 2 infusions four weeks apart
  Interventions: Drug: saline solution

INTERVENTIONS:
Drug: tocilizumab — Le tocilizumab is administered by intravenous infusion at a dose of 8 mg / kg.
  Other Names: ROACTEMRA®
  Arms: tocilizumab
Drug: saline solution — La saline solution is administered by intravenous infusion.
  Other Names: NaCl 0,9 %
  Arms: saline solution

SUMMARY:
Hand osteoarthritis (HOA) which affects the interphalangeal joints and the metacarpophalangeal of the thumb is a common disease, the prevalence of which being about 30 % of the population over than 70. Some forms of HOA are refractory to usual treatments (analgesics, NSAIDs, local injections) and can lead to a high disability. In vitro and in vivo studies showed that IL-6 is involved in the OA process. The aim of the present study is to assess the efficacy of an Interleukin-6-Receptor Inhibitor (tocilizumab) on pain and function in patients with refractory hand OA.

DETAILED DESCRIPTION:
Patient is randomized to receive investigational product or placebo at week 0 and week 4 (1:1)

* arm 1: 2 infusions four weeks apart of tocilizumab 8mg/kg
* arm 2: 2 infusions four weeks apart of saline solution

Follow-up visits are organized at week 6, and then week 8 and week 12.

Primary outcome is the pain as assessed with the VAS at week 6. Secondary outcomes include morning stiffness duration, patient and practitioner global assessments, functional indexes for hand OA, number of painful joints, number of swollen joints.

110 patients is expected to be randomized in 36 months. Each patient sign an informed consent before the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-85
* Hand OA according to the ACR criteria (with recent X-rays of the hands - less than 6 months )
* Symptomatic hand OA lasting more than 3 months (DIP or PIP) despite analgesics and NSAIDs
* OA affecting more than three finger joints (DIP or PIP) (Kellgren and Lawrence equal or more than 2)
* Pain intensity superior to 40 (VAS 0-100 mm) in the last 24 hours
* Not breastfeeding throughout the study and for 150 days after the last infusion
* Negative pregnancy test or effective contraception for women of childbearing age throughout the study and for 150 days after the last infusion or postmenopausal or surgically sterile
* Written informed consent
* Affiliated to health system

Exclusion Criteria:

* Patients having already been treated with an anti-TNF alpha within 6 months
* Patients having already been treated with an Interleukin-6-Receptor Inhibitor
* Hand OA secondary to inflammatory rheumatism
* Existence of painful syndrome of upper limbs likely to interfere with the monitoring of pain (cervicobrachial neuralgia, incapacitating carpal tunnel syndrome, joint disorders of the elbow or shoulder)
* Inflammatory rheumatism
* Psoriasis
* Contraindications to Interleukin-6-Receptor Inhibitor
* Contraindications to acetaminophen
* Anticoagulant (oral) or treatment with heparin at a curative dose
* Surgery scheduled within 6 months following recruitment
* Local injection of a corticosteroid in a symptomatic finger joint during the previous month
* Local injection of hyaluronic acid in a symptomatic finger joint during the prior 6 months
* Treatment with a slow-acting anti-osteoarthritis agent initiated within the previous 3 months
* Treatment with methotrexate, hydrochloroquine, sulfasalazine, colchicine within the last month
* History of symptomatics sigmoiditis or intestinal ulceration
* Oral corticosteroid within 3 days for hydrocortisone or cortisone, within 8 days for prednisone, prednisolone, methylprednisolone or triamcinolone, and within 12 days for betamethasone or dexamethasone
* Psychiatric illness
* Antidepressants initiated or modified within previous month
* Non-controlled diabetes "mellitus"
* Known viral hepatitis B or C, HIV infection
* Current infectious (active or latent tuberculosis)
* Excessive drinking
* Participation in another search
* Lidocain plasters on digital joint within two months

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Change of pain | 6 weeks
  Change of pain between the first infusion (week 0) and 2 weeks after the second infusion (week 6) as assessed on the VAS (0 -100 mm)

SECONDARY OUTCOMES:
Change of pain | weeks 4, 8, 12
  Change of pain between the first infusion (week 0) and 4, 8,12 weeks after the first infusion as assessed on the VAS (0 -100 mm)
Number of painful joints | weeks 4, 6, 8, 12
Number of swollen joints | weeks 4, 6, 8, 12
Overall assessment of disability | weeks 4, 6, 8, 12
  Patient and practitioner global assessments
Morning stiffness duration | weeks 4, 6, 8, 12
Evaluation of the function | weeks 4, 6, 8, 12
  Dreiser's algofunctional index + Functional Cochin hand index

CONTACTS AND LOCATIONS:
Overall Officials: Richette Pascal, MD, PhD, Study Director — Rheumatology department, Lariboisière Hospital
Locations (1):
- Rheumatology department Lariboisiere Hospital, Paris, Île-de-France Region, France